CLINICAL TRIAL: NCT00091715
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Study to Assess the Efficacy, Safety, and Tolerability of Bosentan in Patients With Mildly Symptomatic Pulmonary Arterial Hypertension (PAH)
Brief Title: Efficacy and Safety of Oral Bosentan in Pulmonary Arterial Hypertension Class II
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EARLY; AC-052-364
Record Dates: First submitted 2004-09-16; First posted 2004-09-20 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary arterial hypertension; PAH; PPH; bosentan; early
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension | interventions — Bosentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): 62.5 mg table twice a day for 4 weeks followed by 125 mg tablet twice a day for 6 months followed by an open label period until end of study.
  Interventions: Drug: bosentan
- 2 (Placebo Comparator): placebo for 6 months followed by an open label period
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: bosentan — 65 mg tablet twice a day for 4 weeks followed by 125 mg tablet twice a day until end of study
  Other Names: Tracleer
  Arms: 1
Drug: placebo — placebo for 6 months followed by an open-label period
  Arms: 2

SUMMARY:
The present trial investigates a possible use of oral bosentan, which is currently approved for the treatment of symptoms of pulmonary arterial hypertension (PAH) Class III and IV, to patients suffering from PAH Class II.

ELIGIBILITY:
Inclusion Criteria:

* PAH NYHA Class II
* Significant elevation of mean pulmonary arterial pressure
* Significant elevation of pulmonary vascular resistance at rest
* Limited 6-minute walk distance

Exclusion Criteria:

* PAH secondary to portal hypertension, complex congenital heart disease or reverse shunt
* Restrictive or obstructive lung disease
* Significant vasoreactivity
* Treatments for PAH (within 4 weeks of randomization)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2004-04; Primary Completion 2006-11 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
exercise capacity | Baseline to end of study
cardiac hemodynamics | Baseline to end of study

CONTACTS AND LOCATIONS:
Locations (33):
- United States (6):
  - University of Alabama-Birmingham, Birmingham, Alabama
  - Harbor UCLA Medical Center, Torrance, California
  - Tufts- New England Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - St. Paul University Hospital, Dallas, Texas
- Australia (3):
  - The Prince Charles Hospital, Brisbane
  - Royal Prince Albert Hospital, Camperdown
  - St. Vincent's Hospital, Darlinghurst
- General Hospital of Vienna, Vienna, Austria
- UZ Gasthuisberg, Leuven, Belgium
- Canada (6):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - Halifax Infirmary, Halifax, Nova Scotia
  - Victoria Medical Centre, Hamilton, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Centre de Pneumologie de L'Hospital Laval, Sainte-Foy, Quebec
- Queen Mary Hospital, Hong Kong, China
- Interni klinika VFN, Prague, Czechia
- Marseille-Timone, Marseille, France
- Germany (5):
  - Universitat Greifswald, Greifswald
  - Universitarsklinikum Hamburg-Eppendorf, Hamburg
  - Medizinische Universitatsklinik, Heidelberg
  - Universitatsklinikim Leipzig, Leipzig
  - Klinikum der Universitat Regensburg, Regensburg
- Policlinico S. Orsola-Malpighi, Bologna, Italy
- Netherlands (2):
  - VU Medisch Centrum, Amsterdam
  - University Hospital Maastricht, Maastricht
- Spain (3):
  - Hospital Clinic, Barcelona
  - Hospital Valle d'Hebron, Barcelona
  - Hospital 12 de Octubre, Madrid
- Zurich University Hospital, Zurich, Switzerland
- Papworth Hospital, Cambridge, United Kingdom

REFERENCES:
- [Derived] Galie N, Rubin Lj, Hoeper M, Jansa P, Al-Hiti H, Meyer G, Chiossi E, Kusic-Pajic A, Simonneau G. Treatment of patients with mildly symptomatic pulmonary arterial hypertension with bosentan (EARLY study): a double-blind, randomised controlled trial. Lancet. 2008 Jun 21;371(9630):2093-100. doi: 10.1016/S0140-6736(08)60919-8. PMID 18572079